CLINICAL TRIAL: NCT06735677
Title: Effects of Sexual Health Education During Pregnancy on Sexual Myths, Sexual Function, and Quality of Sexual Life: a Randomized Controlled Study
Brief Title: Sexual Health and Sexual Myths During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Zehra Incedal Sonkaya, Asst. Prof., Amasya University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 182213
Record Dates: First submitted 2024-12-06; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy
Keywords: Sexual myths; reproductive health; sexual attitudes; sexual health education
MeSH Terms: interventions — Sex Education

STUDY DESIGN:
Intervention Model Description: Data collection forms were administered to 100 pregnant women who attended the pregnancy school of a city hospital in a province of Türkiye and agreed to participate in the study. The participants were then randomly assigned by lot into intervention (n=50) and control (n=50) groups. Pregnant women in the intervention group received four training sessions over one month. These sessions covered reproductive health, sexual activity during pregnancy and the postpartum period, personal and sexual hygiene, domestic violence during pregnancy, and misconceptions about pregnancy. Following the completion of the training sessions, the Sexual Quality of Life-Female (SQOL-F) questionnaire and the Female Sexual Function Index (FSFI) were re-administered to all participants for final evaluation. Written informed consent was obtained from all participants before the study commenced. The study was completed with 90 participants (45 in the intervention group and 45 in the control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Education (Experimental): These sessions covered reproductive health, sexual activity during pregnancy and the postpartum period, personal and sexual hygiene, domestic violence during pregnancy, and misconceptions about pregnancy.
  Interventions: Behavioral: sexual health education

INTERVENTIONS:
Behavioral: sexual health education — These sessions covered reproductive health, sexual activity during pregnancy and the postpartum period, personal and sexual hygiene, domestic violence during pregnancy, and misconceptions about pregnancy.

SUMMARY:
The aim of this experimental study is to learn the effects of sexual health education during pregnancy on sexual myths, sexual function and quality of sexual life. The main question it aims to answer is:

Is sexual health education effective in correcting sexual myths? Is sexual health education intervention effective in improving quality of sexual life? Is sexual health education intervention effective in improving sexual function? Participants who received the educational intervention prepared to improve quality of sexual life, sexual myths and sexual function will answer the survey questions after the completion of the training program.

DETAILED DESCRIPTION:
Pregnancy, birth and the postpartum period are important processes in which expectant mothers and fathers experience many physiological, psychological and social changes. Pregnancy is also one of the periods when sexuality is most affected and sexual dysfunctions are commonly seen during this period. Despite the age of information and technology, sexual inexperience or lack of knowledge, growing up in a conservative society, deficiencies in sexual education and false beliefs and myths about sexuality are among the common causes of sexual dysfunction in women. These factors affect couples' attitudes and behaviors regarding sexuality during a sensitive period such as pregnancy, causing couples to experience negativities in their sexual lives.

Sexual dysfunction in women is a complex problem affected by many biological, psychological and individual factors. It is stated that sexual dysfunction in women is a common problem that increases with age and affects 30% to 50% of women, but it is known that its prevalence is quite high among young women.

Sexual life quality can be defined as the individual's perception of their own sexual life in a culture and value system according to their personal goals, expectations, criteria and earnings. Almost all sexual myths consist of negative attitudes such as sexual intercourse during pregnancy being harmful, and these attitudes also negatively affect the quality of sexual life.

By receiving consultancy services on how to have sexual life during pregnancy and obtaining information from the right sources, the prevalence of sexual myths during pregnancy will decrease and the effect on the quality of sexual life during pregnancy will be minimized.

This study aims to provide training to the target group of pregnant women on issues such as reproductive health, changes that may occur due to pregnancy, sexual activity during pregnancy and the postpartum period, and hygiene. The aim of these trainings is to inform pregnant women about sexual health and to increase the quality of their sexual life.

ELIGIBILITY:
Inclusion Criteria:

* At least primary school graduate
* Being in the 18-49 age group
* Being pregnant

Exclusion Criteria:

* Having a condition that prevents communication
* Receiving hospital treatment during the data collection process

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female gender is suitable for participation in the study.
Enrollment: 90 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Sexual Quality of Life-Female | 4 weeks.
  Increase in sexual life quality scores at the end of the training program.
Female Sexual Function Index | 4 weeks.
  Increase in sexual function index scores at the end of the training program.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sütçü İmam University Faculty of Medicine Pregnant School, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No